CLINICAL TRIAL: NCT00900575
Title: Cervical Cancer Detection Using Optical Spectroscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00008173
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; LEEP; colposcopy; Pap smear
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colposcope (Experimental): Patients referred for GYN procedures. Specifically, patients will be referred for Pap smear, colposcope or LEEP. The intervention for this arm is the use of the bench-top, miniature optical spectrometer or trans-vaginal colposcope
  Interventions: Device: Optical Spectroscopy Bench-Top System; Device: Portable Optical Spectrometer; Device: Transvaginal colposcope

INTERVENTIONS:
Device: Optical Spectroscopy Bench-Top System — This device is a bench-top optical spectrometer
Device: Portable Optical Spectrometer — This device is a portable optical spectrometer
Device: Transvaginal colposcope
  Other Names: TVDC; Transvaginal digital colposcope, Pocket colposcope, callascope

SUMMARY:
The objective of the work described in this protocol is to determine the optical signatures of cervical dysplasia using optical technologies.

ELIGIBILITY:
Inclusion Criteria:

* undergoing colposcopy for the diagnosis of cervical cancer
* LEEP for the treatment of cervical cancer in early stages.
* Follow-up Pap smear in surveillance

Exclusion Criteria:

* Women under the age of 18 (minors) will be excluded from this study.
* patients will be excluded if she has had a recent episode of bleeding or preterm labor.
* Subjects who are not competent to give consent will excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2006-05 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Identification of optical signatures of cervical tissue | Day of procedure (less than 10 minutes)
  The primary outcome of this study is the identification of the optical signatures of cervical tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Nimmi Ramanujam, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Chang VT, Cartwright PS, Bean SM, Palmer GM, Bentley RC, Ramanujam N. Quantitative physiology of the precancerous cervix in vivo through optical spectroscopy. Neoplasia. 2009 Apr;11(4):325-32. doi: 10.1593/neo.81386. PMID 19308287
- [Derived] Asiedu MN, Agudogo JS, Dotson ME, Skerrett E, Krieger MS, Lam CT, Agyei D, Amewu J, Asah-Opoku K, Huchko M, Schmitt JW, Samba A, Srofenyoh E, Ramanujam N. A novel speculum-free imaging strategy for visualization of the internal female lower reproductive system. Sci Rep. 2020 Oct 6;10(1):16570. doi: 10.1038/s41598-020-72219-9. PMID 33024146
- See also: PI website to see ongoing research — https://www.globalwomenshealthtechnologies.com/